CLINICAL TRIAL: NCT00239694
Title: Immunogenicity of Pneumococcal Vaccination and Revaccination in Older Adults
Brief Title: PPV: Pneumococcal Polysaccharide Vaccine in Older Adults
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: AG0055
Record Dates: First submitted 2005-10-13; First posted 2005-10-17 (Estimated); Last update posted 2015-08-04 (Estimated); Status verified 2015-07

CONDITIONS: Aging
Keywords: Immune response; Antibody response
MeSH Terms: interventions — Pneumococcal Vaccines; Meningococcal Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Previously vaccinated
  Interventions: Biological: Pneumococcal Vaccine
- 2 (Experimental): Never vaccinated
  Interventions: Biological: Pneumococcal Vaccine; Biological: Meningococcal Vaccine

INTERVENTIONS:
Biological: Pneumococcal Vaccine — One time preventative vaccine
  Other Names: Pneumovax
Biological: Meningococcal Vaccine — One time preventative vaccine
  Other Names: Menomune
  Arms: 2

SUMMARY:
The purpose of this study is to measure how long the improvement in the immune system lasts in older people after they have been vaccinated, and to examine the immune response in older people who get vaccinated a second time.

DETAILED DESCRIPTION:
Streptococcus pneumonia is the leading cause of pneumonia the United States, estimated to cause at least 500,000 cases annually and 40,000 deaths. Interest in expanding pneumococcal vaccine administration has arisen with the increased prevalence of antibiotic-resistant S. pneumoniae, increasing numbers of people living with chronic medical conditions, and the aging population.

Extensive studies on vaccine response in older persons have been performed over the past 25 years. However, a number of issues hindered the assessment of vaccine response in older people. Recent studies indicate most healthy older people develop an initial antibody response to vaccination similar to younger cohorts, although antibody response to some serotypes may be less. Limited data suggest functional antibody will develop at least initially after vaccination in older recipients. There are no published reports describing the duration of antibody response or antibody function after revaccination in older patients.

It is difficult to predict the revaccination response and, for those with elevated pre-revaccination antibody, there may be no response to revaccination, or even a lowering of absolute antibody level. Accordingly, a well-controlled revaccination protocol in which older patients with defined vaccine history and known pre-revaccination antibody level are studied for quantitative and qualitative antibody response to revaccination is sorely needed.

The hypotheses for this study are:

1. Specific antipneumococcal antibody will remain above prevaccination level in the serum of healthy older people for up to ten years after PPV.
2. Healthy older people will have a prompt and robust vaccine response to primary vaccination with PPV.
3. The existence of antipneumococcal antibody in healthy older people who had been vaccinated with PPV >5 years previously will not be associated with more pronounced or frequent adverse events or a reduced vaccine response rate.
4. The effect of advanced age will account for a reduced vaccine response.

Volunteers in the Baltimore Longitudinal Study of Aging (BLSA) will be asked to participate in this retrospective/prospective analysis. Two pools of participants will be recruited. The first group (Group I) will be 65 years and older who had received PPV five or more years earlier, and the second (Group II) will be decade and gender matched individuals with no prior exposure to PPV. These groups will be matched as closely as possible.

All volunteers (Groups I and II) will receive the same vaccines. In one arm they will receive PPV (for group I this will be revaccination and for group II this will be primary vaccination). In the other arm they will receive Meningococcal Polysaccharide Vaccine (MPV) (primary vaccination for both groups I and II).

Blood samples will be drawn before and after vaccination on day 0 (the day of vaccination), on day 28, and at 6 months following vaccination. Approximately six months after the last vaccination participants will be asked to complete a brief medical history update, either by telephone, by mail, or during their regularly scheduled BLSA visit. This update will continue to be performed every six months for the duration of the study.

ELIGIBILITY:
Inclusion Criteria:

* Enrolled in the BLSA with at least 2 stored blood samples post vaccination
* 65 years old or older
* Previously vaccinated with Pneumovax at least 5 years ago or never vaccinated
* Willing to receive vaccination with pneumococcal and meningococcal injection
* Able to provide informed consent
* Has never received a meningococcal vaccine

Exclusion Criteria:

* Hypersensitivity to the pneumococcal or meningococcal vaccine
* Ever received the Meningococcal vaccine
* History of non-skin cancer
* History of myeloproliferative disorder
* History of HIV
* Received a Bone Marrow Transplant
* Taking prednisone (more than 5 mg/day) or other immunosuppressive medication
* Evidence of severe liver or renal disease (serum creatine >2.0 mg/dL or Total Bilirubin >2.0

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 100 (Actual)
Dates: Start 2001-04; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Pre and post vaccination (groups I and II) serum samples | Day 0, day 28, and 6 months following vaccination and days on each BLSA site visit

CONTACTS AND LOCATIONS:
Overall Officials: Dan L. Longo, MD, Principal Investigator — Scientific Director, National Insitute on Aging
Locations (1):
- National Institute on Aging, Baltimore, Maryland, United States

REFERENCES:
- [Background] Hedlund J, Ortqvist A, Konradsen HB, Kalin M. Recurrence of pneumonia in relation to the antibody response after pneumococcal vaccination in middle-aged and elderly adults. Scand J Infect Dis. 2000;32(3):281-6. doi: 10.1080/00365540050165929. PMID 10879599
- [Background] Musher DM, Luchi MJ, Watson DA, Hamilton R, Baughn RE. Pneumococcal polysaccharide vaccine in young adults and older bronchitics: determination of IgG responses by ELISA and the effect of adsorption of serum with non-type-specific cell wall polysaccharide. J Infect Dis. 1990 Apr;161(4):728-35. doi: 10.1093/infdis/161.4.728. PMID 2319166
- [Background] Hilleman MR, Carlson AJ Jr, McLean AA, Vella PP, Weibel RE, Woodhour AF. Streptococcus pneumoniae polysaccharide vaccine: age and dose responses, safety, persistence of antibody, revaccination, and simultaneous administration of pneumococcal and influenza vaccines. Rev Infect Dis. 1981 Mar-Apr;3 Suppl:S31-42. doi: 10.1093/clinids/3.supplement_1.s31. PMID 7025159